CLINICAL TRIAL: NCT03603912
Title: Upstream Targeting for the Prevention of Atrial Fibrillation: Targeting Risk Interventions and Metformin for Atrial Fibrillation (TRIM-AF)
Brief Title: Targeting Risk Interventions and Metformin for Atrial Fibrillation (TRIM-AF)
Acronym: TRIM-AF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mina Chung, MD (Other)
Collaborators: American Heart Association (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Mina Chung, MD, Principal Investigator, Professor of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 18-757
Record Dates: First submitted 2018-07-12; First posted 2018-07-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Control (No Intervention): Written educational literature on healthy eating and exercise guideline
- Metformin (Experimental): Metformin ER up to 750 mg twice daily
  Interventions: Drug: Metformin
- Lifestyle/Risk Factor Modification (Experimental): Lifestyle/Risk Factor Modification (LRFM): Diet/nutrition, exercise, and risk factor modification
  Interventions: Behavioral: Lifestyle/Risk Factor Modification
- Metformin + LRFM (Experimental): Metformin ER up to 750 mg twice daily + Lifestyle/Risk Factor Modification (LRFM) diet/nutrition, exercise, and risk factor modification
  Interventions: Drug: Metformin; Behavioral: Lifestyle/Risk Factor Modification
- No Atrial Fibrillation (No Intervention): Written educational literature on healthy eating and exercise guideline

INTERVENTIONS:
Drug: Metformin — Metformin ER 500 mg daily, titrated at 1 month intervals to 500 mg twice daily, then 750 mg twice daily, as tolerated, for 2 years.
  Other Names: Metformin HCL
  Arms: Metformin; Metformin + LRFM
Behavioral: Lifestyle/Risk Factor Modification — Diet/nutrition counseling and exercise prescription with follow-up visits, sleep apnea screening and treatment if detected, optimization of guideline-directed medical therapies for hypertension, coronary artery disease (CAD), hyperlipidemia and heart failure (HF).
  Other Names: LRFM
  Arms: Lifestyle/Risk Factor Modification; Metformin + LRFM

SUMMARY:
Prospective randomized open-label blinded endpoint (PROBE) 2x2 factorial study of metformin extended release up to 750 mg BID and lifestyle and risk factor modification (LRFM) in CIED patients with at least 1 ≥5 minute episode of AF over the prior 3 months. Randomization will be stratified by pacemaker vs. ICD and rhythm at enrollment (sinus rhythm/atrial paced vs. AF).

DETAILED DESCRIPTION:
The purpose of this study is to perform a prospective, randomized study for the reduction of atrial fibrillation (AF) burden and progression, targeting metabolic upstream therapies. The study aims to determine if metformin and/or lifestyle/risk factor modifications reduce AF burden and progression. A secondary aim will attempt to determine clinical, genomic, and biomarker predictors of AF progression that can be used to personalize upstream therapies. This is a prospective randomized open-label blinded endpoint (PROBE) 2x2 factorial study of metformin extended release up to 750 mg twice daily and lifestyle and risk factor modification (LRFM) in patients with implanted pacemakers or defibrillators with atrial leads and at least 1 ≥5 minute episode of AF over the prior 3 months.

ELIGIBILITY:
TRIM-AF Cohorts

Inclusion Criteria:

1. Permanent pacemaker or implantable cardioverter-defibrillator (ICD) (with or without cardiac resynchronization therapy (CRT) with an implanted atrial lead capable of providing AF diagnostics and remote monitoring.
2. Paroxysmal AF, or persistent AF with plans for conversion.
3. AF on cardiac implantable electrical device (CIED) over the past 3 months with at least 1 episode lasting ≥5 minutes.
4. If on an antiarrhythmic drug, then on a stable regimen for the past 3 months.

Exclusion Criteria:

1. Permanent AF with no plans to convert to sinus rhythm.
2. If in persistent AF, current episode >12 months in duration (current long-standing persistent AF)
3. NYHA Functional Class IV heart failure
4. On metformin or other pharmacologic therapy for diabetes mellitus.
5. Use of anti-retroviral protease inhibitors (e.g. ombitasvir, paritaprevir, ritonavir, dasabuvir) or topiramate.
6. Known sensitivity to metformin
7. Moderate renal disease (eGFR <45 ml/min/1.73 m2)
8. Significant alcohol use (average >2 drinks/day)
9. Hepatic dysfunction - bilirubin >1.5x ULN, unless due to Gilbert's syndrome
10. Planned antiarrhythmic (class I or III) drug change, AF ablation/PVI procedure or cardiac surgery over the first 3 mos of the study
11. AF ablation/PVI procedure performed in the past 6 months
12. Device changed or implanted in the past 3 months
13. For patients on dofetilide with a pacemaker, QTc >490 ms if QRS duration is </=100 ms. If QRS duration is >100 ms, adjusted QTc >490 ms. Adjusted QTc = QTc - (QRS duration - 100 ms).
14. Women who are pregnant, breast-feeding or of child-bearing potential and not willing or able to use an acceptable form of contraception.
15. Participants considered by the investigator to be unsuitable for the study for any of the following reasons: Not agreeable for treatment with metformin or anticipated to have poor compliance on study drug treatment; inability to follow diet or exercise instructions; unwilling to attend study follow-up visits
16. Life expectancy less than 2 years due to concomitant disease.
17. Age <18 years old.

TRIM - No AF Cohort

Inclusion Criteria:

1. Permanent pacemaker or ICD (with or without CRT) with an implanted atrial lead capable of providing AF diagnostics and remote monitoring.
2. No AF on CIED over the past 6 months.
3. No history of AF.
4. Age >/=18 years old.

Exclusion Criteria:

1. History of AF.
2. NYHA Functional Class IV heart failure
3. On metformin or other pharmacologic therapy for diabetes mellitus.
4. Use of anti-retroviral protease inhibitors (e.g. ombitasvir, paritaprevir, ritonavir, dasabuvir) or topiramate.
5. Moderate renal disease (eGFR <45 ml/min/1.73 m2)
6. Significant alcohol use (average >2 drinks/day)
7. Hepatic dysfunction - bilirubin >1.5x ULN, unless due to Gilbert's syndrome
8. Planned antiarrhythmic (class I or III) drug change, cardiac surgery over the first 3 mos of the study
9. Device changed or implanted in the past 3 months
10. For patients on dofetilide with a pacemaker, QTc >490 ms if QRS duration is </=100 ms. If QRS duration is >100 ms, adjusted QTc >490 ms. Adjusted QTc = QTc - (QRS duration - 100 ms).
11. Women who are pregnant, breast-feeding or of child-bearing potential and not willing or able to use an acceptable form of contraception.
12. Participants considered by the investigator to be unsuitable for the study for any of the following reasons: Not agreeable for treatment with metformin or anticipated to have poor compliance on study drug treatment; inability to follow diet or exercise instructions; unwilling to attend study follow-up visits
13. Life expectancy less than 2 years due to concomitant disease.
14. Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in AF burden | 1 year
  Composite of change from baseline to 1 year of average daily AF burden % after a 3 month blanking period and survival at 1 year.

SECONDARY OUTCOMES:
Total time of AF/3 mos | 3 months, 1 year, 2 years
  Total time of AF per 3 month period
Average %time in AF/day | 3 months, 1 year, 2 years
  Average percent time in AF/day
%change in average AF time/day | Baseline to 3 months, 1 year, 2 years
  Percent change in average AF time/day from baseline
Number of days of AF | 3 months, 1 year, 2 years
  Number of days of AF over the time period
Number of AF episodes/month | 3 months, 1 year, 2 years
  Number of AF episodes/month over the time period
Longest duration of AF at each 3 mo. period | 3 months, 1 year, 2 years
  Longest duration at each 3 mo. period over the time period
Change in AF burden without blanking period | 1 year
  Composite of change from baseline to 1 year of average daily AF burden % and survival at 1 year.
AF density | 1 year, 2 years
  a measure of AF temporal aggregation, calculated using daily AF burden time over the study period
Time to next AF and to persistent AF | Up to 2 years
  Time to next AF and to persistent AF with and without a 3 mo. blanking period
Incidence of Persistent AF | 3 months, 1 year, 2 years
  Development of persistent AF over the study period
Cardioversion for AF | 3 months, 1 year, 2 years
  Electrical cardioversion procedures over the study period
AF ablation/pulmonary vein isolation (PVI) for increase in burden or persistent AF | 3 months, 1 year, 2 years
  Occurrence of AF ablation/PVI procedures over the study period.
Change of antiarrhythmic drug | 3 months, 1 year, 2 years
  Change or new initiation of class I or III antiarrhythmic drug over the study period.
Change in Atrial Fibrillation Symptom Score (AFSS) | Baseline, 1 year, 2 years
  Changes in Atrial Fibrillation Symptom Score (AFSS) from baseline - Global well-being (1-10), AF duration (1-8, lower denotes longer duration AF), AF severity (1-10, higher denotes more severe AF), ER visits (0-7), Hospitalizations (0-7), Specialist visits (0-7)
Change in Short Form-36 (SF-36) scores | Baseline, 1 year, 2 years
  Change in SF-36 scores from baseline. SF-36 has 8 scaled scores; scores are weighted sums of the questions in each section. Scores range from 0-100 with lower scores indicating more disability, higher scores indicating less disability. Sections are: Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Change in physical assessment questionnaire scores: Rapid Assessment of Physical Activity (RAPA) | Baseline, 1 year, 2 years
  Change in physical assessment questionnaire score from baseline. RAPA 1 Aerobic score 1-7, high more active. RAPA 2 Strength & Flexibility score 0-3 (higher more strength and flexibility)
Change in GPCOG questionnaire score | Baseline, 1 year, 2 years
  Change in General Practitioner assessment of Cognition (GPCOG) questionnaire score from baseline. Step 1: Score 0-4 Cognitive impairment is indicated; 5-8 More information required; 9 No significant cognitive impairment
Change in weight | baseline, 1 year, 2 years
  Change in weight (pounds) from baseline
Change in body fat composition | baseline, 1 year, 2 years
  Change in body fat composition (%) from baseline.
Change in BMI | Baseline, 1 year, 2 years
  Change in body mass index (BMI, kg/m2) from baseline (calculated from weight, height)
Change in waist/hip ratio | Baseline, 1 year, 2 years
  Change in waist/hip ratio from baseline
Change in HbA1c | Baseline, 1 year, 2 years
  Change in HbA1c (%) from baseline
Change in total cholesterol | Baseline, 1 year, 2 years
  Change in total cholesterol from baseline
Change in LDL | Baseline, 1 year, 2 years
  Change in LDL from baseline
Change in HDL | Baseline, 1 year, 2 years
  Change in HDL from baseline
Change in triglycerides | Baseline, 1 year, 2 years
  Change in triglycerides from baseline
Change in Homeostatic Model Assessment - Insulin Resistance (HOMA-IR) | Baseline, 1 year, 2 years
  Change in HOMA-IR from baseline (calculated from fasting blood sugar and insulin)
Composite Major Adverse Cardiovascular Events (MACE) | 1 year, 2 years
  Composite incidence of cardiovascular death, nonfatal stroke, nonfatal myocardial infarction
All-cause mortality | 1 year, 2 years
  Incidence of all-cause death
Stroke | 1 year, 2 years
  Incidence of stroke
Transient ischemic attack | 1 year, 2 years
  Incidence of transient ischemic attack
Activity by implanted device | 3 months, 1 year, 2 years
  Daily activity as measured by the sensors in the implanted pacemaker or defibrillator device (hours/day)

CONTACTS AND LOCATIONS:
Overall Officials: Mina K Chung, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wass SY, Barnard J, Kim HS, Sun H, Telfer W, Schilling T, Barzilai B, Bruemmer D, Cho L, Huang J, Hussein A, Kashyap SR, Laffin L, Mehra R, Moravec C, Saliba W, Sanders P, Nissen S, Varma N, Smith J, Van Wagoner D, Chung MK. Upstream targeting for the prevention of atrial fibrillation: Targeting Risk Interventions and Metformin for Atrial Fibrillation (TRIM-AF)-rationale and study design. J Interv Card Electrophysiol. 2025 Jan;68(1):9-19. doi: 10.1007/s10840-024-01955-z. Epub 2024 Dec 13. PMID 39671157